CLINICAL TRIAL: NCT01253382
Title: A 3-Part Study to Evaluate the Pharmacokinetics, Safety, and Efficacy of Subcutaneous Ecallantide in Prepubertal Paediatric Patients Experiencing Acute Attacks of Hereditary Angioedema (HAE)
Brief Title: Study to Evaluate Ecallantide in Paediatric Patients With Acute Attacks of Hereditary Angioedema
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DX-88/26; 2010-022716-39 (EudraCT Number)
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Hereditary Angioedema (HAE)
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — ecallantide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ecallantide (Active Comparator)
  Interventions: Biological: ecallantide
- placebo (Placebo Comparator): phosphate buffered saline
  Interventions: Biological: ecallantide

INTERVENTIONS:
Biological: ecallantide — 10 - 30mg subcutaneous injection.

SUMMARY:
The primary objective of this study is:

* assess the safety and tolerability of ecallantide in paediatric patients for acute attacks of HAE

The secondary objectives are:

* evaluate the pharmacokinetic profile of ecallantide in paediatric patients treated for acute attacks of HAE
* assess the efficacy of ecallantide in paediatric patients treated for moderate to severe acute attacks of HAE

ELIGIBILITY:
Inclusion Criteria:

1. Male or female from 2 years of age and prepubertal
2. Physician diagnosis and history of HAE (Type I or II) including laboratory results showing C1-1NH activity below the lower limit of normal or up to 15% above the lower limit of the normal range
3. Present at the site with moderate to severe signs and symptoms of an acute attack of HAE within 8 hours of recognition of the onset of the attack. Spontaneous resolution of the attack must not have begun before the administration of study drug.
4. Must have signed informed consent by parent or caregiver.

Exclusion Criteria:

1. <2 years of age or have reached puberty
2. Received treatment with ecallantide within previous 72 hours
3. Received an investigational drug or device, other than ecallantide, within 30 days prior to the screening visit
4. Pharyngeal/laryngeal symptoms
5. Mild attacks including mild edema of the extremities and mild abdominal attacks
6. Are unable or unwilling to give informed consent (parent or caregiver)
7. Any other condition that, in the opinion of the investigator, may compromise the safety or compliance of the patient or would preclude the patient from successful completion of the study

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2015-04-01 (Estimated)

PRIMARY OUTCOMES:
safety and tolerability of ecallantide | 4 years

SECONDARY OUTCOMES:
evaluate the PK profile of ecallantide | 4 years
assess the efficacy of ecallantide | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda